CLINICAL TRIAL: NCT05304442
Title: Intravenous Ferric Derisomaltose for Moderate to Severe Anemia Due to Uterine Bleeding in the Emergency Department: a Randomized Trial
Brief Title: IV Iron Trial for Anemia Related to Uterine Bleeding in Female Patients Presenting to the Emergency Department
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Pharmacosmos Therapeutics, Inc. (Unknown)
Responsible Party: Principal Investigator, Stephen Boone MD, Assistant Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-49444
Record Dates: First submitted 2022-03-22; First posted 2022-03-31 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Anemia, Iron Deficiency; Uterine Bleeding
Keywords: IV Iron; Emergency Department; Iron Deficiency Anemia; Uterine Bleeding
MeSH Terms: conditions — Anemia, Iron-Deficiency; Uterine Hemorrhage; Emergencies | interventions — ferric derisomaltose; ferrous sulfate

STUDY DESIGN:
Intervention Model Description: Randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intravenous Ferric Derisomaltose (Experimental): One single dose of ferric derisomaltose, 1000 mg Intravenous over at least 20 minutes.
  Interventions: Drug: Ferric Derisomaltose 1000 Mg in 10 mL INTRAVENOUS SOLUTION [Monoferric]
- Oral Iron (Active Comparator): ferrous sulfate 65 mg once daily for 42 days.
  Interventions: Drug: Ferrous Sulfate 65 mg elemental iron (325 mg tablets)

INTERVENTIONS:
Drug: Ferric Derisomaltose 1000 Mg in 10 mL INTRAVENOUS SOLUTION [Monoferric] — Single Dose of IV Iron
  Arms: Intravenous Ferric Derisomaltose
Drug: Ferrous Sulfate 65 mg elemental iron (325 mg tablets) — Once daily by mouth for 42 days
  Arms: Oral Iron

SUMMARY:
The primary aim of this randomized trial is to assess the efficacy of IV Ferric Derisomaltose vs Oral Iron in the management of women with severe Iron Deficiency Anemia due to Uterine Bleeding in the emergency department.

DETAILED DESCRIPTION:
Iron deficiency anemia (IDA) is the most common hematologic disorder in the United States and worldwide. Patients with moderate to severe anemia often present to the acute care setting for initial assessment and evaluation; women with abnormal uterine bleeding are among those at highest risk. Guidelines on management of this common condition in the emergency department (ED) are lacking.

Although IDA is commonly encountered in the ED, there is a paucity of literature addressing optimal management in this setting. Intravenous (IV) iron therapy is infrequently used in the ED despite evidence of safety and superiority to oral iron therapy in other acute care settings. Furthermore, red blood cell (RBC) transfusions may be over-utilized in hemodynamically stable patients with IDA, potentially increasing risk for transfusion reactions, infection, and allo-antibody formation among other adverse outcomes. Improved treatment of iron deficiency may reduce the need for subsequent RBC transfusions. Compared with oral iron, treatment with intravenous iron may result in improved adherence, fewer health care visits, more rapid correction of IDA, and overall improvement in quality of life.

Historically, older formulations of IV Iron, namely high-molecular weight iron dextran (HMWID), were associated with unacceptably high rates of severe allergic reactions and/or required multiple doses to replete iron stores. However, newer formulations of IV iron are not only extremely safe, but can also be administered as a single "total dose infusion" over a very short time period. These newer forms of IV iron include ferric carboxymaltose, low-molecular weight iron dextran, ferumoxytol, and ferric derisomaltose. When excluding HMWID, a meta-analysis of 97 RCTs found that there was no increase in the risk of serious adverse events (SAE's) with IV iron compared with control and no increased risk of systemic infection.

A large retrospective, "before and after" study conducted in an Italian Emergency Department demonstrated that implementation of Patient Blood Management protocols, including the use of IV iron in the emergency department, resulted in a substantial reduction in red blood cell transfusions, hospitalization, re-transfusion, length of stay and costs. Similar conclusions were reached in smaller studies by Motta et al and Khadadah et al.

The investigators recently published a retrospective cohort study examining current emergency department practices in the evaluation and management of IDA in the target population for the proposed trial. The results of this cohort study revealed that women with AUB and severe anemia are frequently seen in the Ben Taub Emergency Department, that red blood cell transfusions are commonly administered, and that IV iron is infrequently (or never) used in the ED setting. Furthermore, unplanned return visits and recurrent transfusions were common.

ELIGIBILITY:
Inclusion Criteria:

* Sub-acute or chronic uterine blood loss;
* Moderate to Severe Anemia, defined as Hgb less than or equal to 9.0 g/dl;
* Iron deficiency: Serum ferritin less than or equal to 30 ng/mL;
* Eligible for discharge from the ED following treatment;
* Patient able to return for planned follow-up visits at 3 and 6 weeks;
* Patient able to be reached by telephone;
* Willing and able to provide consent for participation.

Exclusion Criteria:

* Patient requiring hospitalization for any reason;
* Pregnant or nursing;
* Incarcerated/Prisoner;
* Weight < 50 kg;
* History of hypersensitivity reactions, as specified, known hypersensitivity to any formulation of parenteral iron;
* History of any anaphylactic allergy;
* Recent receipt of IV iron, erythropoiesis-stimulating agents;
* Erythropoiesis-stimulating agent use within 8 weeks prior to ED visit;
* Parenteral iron within 4 weeks prior to ED visit;
* Scheduled/planned use of parenteral iron or ESA during study period;
* Receipt of blood transfusion at index visit;
* Planned elective major surgery during study period;
* Other current or recent hematologic therapy, as specified;
* Current or planned use of antithrombotic therapy (antiplatelet agents or anticoagulants) within study period (Non-aspirin NSAIDs are NOT a contraindication);
* Known bleeding disorder platelets < 100,000';
* Other significant underlying comorbidity, as specified:
* Active rheumatologic disease, or rheumatologist disease requiring treatment, such as rheumatoid arthritis, systemic lupus erythematosus, or mixed connective tissue disease;
* Acute heart failure or NYHA II-IV chronic heart failure;
* Inflammatory bowel disease;
* Cirrhosis or Decompensated liver disease;
* Chronic kidney disease, stage III or greater (eGFR < 60);
* Current Systemic Infection (e.g. pneumonia, pelvic inflammatory disease, pyelonephritis). *Cystitis or cervicitis is NOT an exclusion
* Any other medical or surgical condition that in the opinion of the treating physician may result in patient being unsuitable for trial participation

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-09-15 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
mean change in hemoglobin concentration | 3 weeks
  participants will have increased hemoglobin concentrations

SECONDARY OUTCOMES:
mean change in hemoglobin concentration | 6 weeks
  participants will have increased hemoglobin concentrations

OTHER OUTCOMES:
mean change in ferritin | 3 weeks
  participants will have increased ferritin
mean change in ferritin | 6 weeks
  participants will have increased ferritin
median number of transfusions | 6 weeks
  compare between the two arms
median number of return Emergency Department visits | 6 weeks
  compare between the two arms
adverse events | 6 weeks
  compare between the two arms

CONTACTS AND LOCATIONS:
Locations (1):
- Ben Taub Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferrer-Barcelo L, Sanchis Artero L, Sempere Garcia-Arguelles J, Canelles Gamir P, P Gisbert J, Ferrer-Arranz LM, Monzo Gallego A, Plana Campos L, Huguet Malaves JM, Lujan Sanchis M, Ruiz Sanchez L, Barcelo Cerda S, Medina Chulia E. Randomised clinical trial: intravenous vs oral iron for the treatment of anaemia after acute gastrointestinal bleeding. Aliment Pharmacol Ther. 2019 Aug;50(3):258-268. doi: 10.1111/apt.15327. Epub 2019 Jun 14. PMID 31197861
- [Background] Sultan P, Bampoe S, Shah R, Guo N, Estes J, Stave C, Goodnough LT, Halpern S, Butwick AJ. Oral vs intravenous iron therapy for postpartum anemia: a systematic review and meta-analysis. Am J Obstet Gynecol. 2019 Jul;221(1):19-29.e3. doi: 10.1016/j.ajog.2018.12.016. Epub 2018 Dec 19. PMID 30578747
- [Background] Quintana-Diaz M, Fabra-Cadenas S, Gomez-Ramirez S, Martinez-Virto A, Garcia-Erce JA, Munoz M. A fast-track anaemia clinic in the Emergency Department: feasibility and efficacy of intravenous iron administration for treating sub-acute iron deficiency anaemia. Blood Transfus. 2016 Mar;14(2):126-33. doi: 10.2450/2015.0176-15. Epub 2015 Nov 19. PMID 26674819
- [Background] Beverina I, Razionale G, Ranzini M, Aloni A, Finazzi S, Brando B. Early intravenous iron administration in the Emergency Department reduces red blood cell unit transfusion, hospitalisation, re-transfusion, length of stay and costs. Blood Transfus. 2020 Mar;18(2):106-116. doi: 10.2450/2019.0248-19. Epub 2019 Dec 17. PMID 31855149
- [Background] Motta I, Mantovan G, Consonni D, Brambilla AM, Materia M, Porzio M, Migone De Amicis M, Montano N, Cappellini MD. Treatment with ferric carboxymaltose in stable patients with severe iron deficiency anemia in the emergency department. Intern Emerg Med. 2020 Jun;15(4):629-634. doi: 10.1007/s11739-019-02223-z. Epub 2019 Nov 9. PMID 31707563
- [Background] Khadadah F, Callum J, Shelton D, Lin Y. Improving quality of care for patients with iron deficiency anemia presenting to the emergency department. Transfusion. 2018 Aug;58(8):1902-1908. doi: 10.1111/trf.14626. Epub 2018 Apr 17. PMID 29664169
- [Background] Boone S, Peacock WF, Ordonez E, Powers JM. Management of Nonpregnant Women Presenting to the Emergency Department With Iron Deficiency Anemia Caused by Uterine Blood Loss: A Retrospective Cohort Study. J Emerg Med. 2020 Sep;59(3):348-356. doi: 10.1016/j.jemermed.2020.05.006. Epub 2020 Jun 24. PMID 32593579
- [Background] Achebe M, DeLoughery TG. Clinical data for intravenous iron - debunking the hype around hypersensitivity. Transfusion. 2020 Jun;60(6):1154-1159. doi: 10.1111/trf.15837. Epub 2020 Jun 1. PMID 32479668